CLINICAL TRIAL: NCT00642291
Title: An Open-Label Study of a Once Daily Dose of Emtricitabine in Combination With Other Antiretroviral Agents in HIV Infected Pediatric Subjects
Brief Title: An Open-Label Study of Emtricitabine in Combination With Other Antiretroviral Agents in HIV Infected Pediatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Elsa Mondou, MD, Senior Director of Clinical Research, Gilead Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FTC-211
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections
Keywords: Emtricitabine; Pediatric; HIV-1; Treatment of HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment naive pediatric patients (Group 1: ages 3 to 24 months)were to receive emtricitabine (6mg/kg QD; max 200 mg QD) plus stavudine 1 mg/kg BID (if <30kg)plus lopinavir/ritonavir (12/3 mg/kg BID if >=7 to <15kg; 10/2.5 mg/kg BID if >=15 to <=40 kg)
  Interventions: Drug: Emtricitabine
- 2 (Experimental): Treatment naive or experienced pediatric patients (Group 2: ages 7 to 12 years; Group 3: ages 13-17 years) received emtricitabine (6 mg/kg QD, up to 200 mg QD capsule formulation or up to 240 mg QD using the oral solution) plus didanosine (240 mg/m2 up to 400 mg QD) plus efavirenz (up to 600 mg QD capsule formulation or up to 720 mg QD using the oral solution).
  Interventions: Drug: Emtricitabine

INTERVENTIONS:
Drug: Emtricitabine — emtricitabine (6mg/kg QD; max 200 mg QD) plus stavudine 1 mg/kg BID (if <30kg)plus lopinavir/ritonavir (12/3 mg/kg BID if >=7 to <15kg; 10/2.5 mg/kg BID if >=15 to <=40 kg)
  Other Names: FTC
  Arms: 1
Drug: Emtricitabine — emtricitabine (6 mg/kg QD, up to 200 mg QD capsule formulation or up to 240 mg QD using the oral solution) plus didanosine (240 mg/m2 up to 400 mg QD) plus efavirenz (up to 600 mg QD capsule formulation or up to 720 mg QD using the oral solution).
  Other Names: FTC
  Arms: 2

SUMMARY:
To obtain safety and efficacy data for antiretroviral regimens containing emtricitabine in HIV-1 infected pediatric subjects. To determine emtricitabine concentrations in HIV-1 infected pediatric subjects and, if necessary, to refine the dose of emtricitabine to achieve concentrations comparable to those in adults given 200 mg emtricitabine once-daily.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 3 to 24 months old or from 7 to 17 years old. (Note: This criterion was based on the subject's age at Baseline [Day 1].)
* Documented evidence of HIV-1 infection. (Note: HIV-1 infection had to be confirmed by two positive results obtained in any of the following:
* at any age: HIV culture, HIV DNA PCR, or plasma HIV RNA of >= 10,000 copies/mL;
* age > 4 weeks: neutralizable HIV p24 antigen; or
* age > 18 months: licensed ELISA with confirmatory Western blot.)
* Body weight > 2.5 kg (>5.5 lb).
* Either ART-naïve or ART-experienced, as defined below:
* ART-naïve: no prior exposure to any ART (with the exception of <= 56 cumulative days of perinatal prophylactic treatment for the prevention of maternal-to-child transmission or <=6 weeks of cumulative postnatal treatment with ZDV monotherapy) and a Screening plasma HIV-1 RNA level of >= 5,000 copies/mL and, in children aged >= 7 years old, a plasma HIV-1 RNA of <= 600,000 copies/mL.

OR

* ART-experienced: no previous treatment with an ART regimen(s) that included either lamivudine and/or an NNRTI and a Screening plasma HIV-1 RNA level of <= 600,000 copies/mL.
* Absolute CD4+ cell count of >= 200 cells/mm3.
* Subjects whose parent or other legal guardian provided written informed consent to participate in the study.
* Female subjects of childbearing potential (i.e., post-pubertal) with a negative serum beta human chorionic gonadotropin (Beta-HCG) test at Screening that was confirmed by a negative urine pregnancy test at Baseline, prior to administration of the first dose of emtricitabine.
* If sexually active and/or of childbearing potential, the subject (male and female) had to be willing to use an effective method of contraception while enrolled in the study and for a period of at least 1 month after the last dose of emtricitabine

Exclusion Criteria:

* Either the subject or the subject's parent or other legal guardian was unable to adhere to the child's dosing schedule and protocol evaluations.
* Female subjects who were pregnant or who were breastfeeding.
* Treatment within 30 days prior to Baseline with an investigational drug, agent, and/or vaccine (with the exception of investigational formulations of approved drugs) unless prior approved by both the investigator and sponsor.
* Subjects who required the concomitant use of: (a) immunomodulators (with the exception of immune globulin and colony stimulating factors); (b) investigational drug,agent, and/or vaccines (with the exception of investigational formulations of approved drugs; and/or (c) any medication that was contra-indicated for any protocol-prescribed background medication, unless pre-approved by both the investigator and sponsor.
* Subjects with any of the following laboratory parameters at Screening:

  1. Hemoglobin >= Grade 3 toxicity;
  2. Absolute neutrophil count ≥ Grade 2 toxicity (assessed without Neupogen [filgrastim, G-CSF]);
  3. Platelet count >= Grade 2 toxicity;
  4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >= Grade 2 toxicity;(Note: Re-screening was NOT allowed for an exclusionary AST or ALT value, unless acute viral hepatitis was documented and the elevated ALT and/or AST demonstrated complete resolution with no exclusionary amylase or lipase value.)
  5. Serum creatinine >= Grade 2 toxicity;
  6. Total bilirubin >= Grade 2 toxicity (other than for Gilbert's syndrome); and
  7. Pancreatic amylase or total amylase plus lipase >= Grade 2 toxicity. (Note: Re-screening was NOT allowed for exclusionary amylase or lipase values.)
* Subjects with any other clinical or laboratory abnormality of >= Grade 3 toxicity (using age-specific toxicity grading scales for children < 13 years old and >= 13 years old at Screening unless pre-approved by the investigator and sponsor.
* Subjects with >= Grade 2 peripheral neuropathy at Screening or with a significant history of peripheral neuropathy.
* Subjects with malabsorption or severe chronic diarrhea (>= Grade 2) within 30 days before Screening, or subjects who were unable to consume adequate oral intake (defined as the inability to eat >= 1 meal(s) a day or to have 3 feedings a day for young infants) because of chronic nausea, emesis, or abdominal or esophageal discomfort.
* Subjects with an acute and serious medical event within 30 days prior to Screening unless pre-approved by the investigator and sponsor. (Note: Acute treatment must have been completed for >= 14 days prior to Baseline.)
* Subjects with an AIDS-defining opportunistic infection within 12 months prior to Screening.
* Life expectancy < 12 months.
* Subjects currently being treated for active tuberculosis.
* Subjects with a history of acute or chronic (clinical or biological) pancreatitis (regardless of their serum amylase levels).
* Any other condition or set of circumstances, which, in the opinion of the investigator or sponsor, could have interfered with the subject's ability to comply with the dosing schedule and complete the study evaluations.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2002-11; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint was tolerability failure (A patient was classified as a tolerability failure if (s)he had any adverse event or laboratory toxicity that lead to the permanent discontinuation of emtricitabine | Week 48
The primary efficacy endpoint was defined as the suppression of plasma HIV-1 RNA levels below 50 copies/mL at Week 48 | Week 48

SECONDARY OUTCOMES:
Time to loss of virological response (TLOVR) | Week 48
plasma HIV-1 RNA change from baseline | Week 48
proportion of patients with plasma HIV-1 RNA below 400 copies/mL | Week 48
CD4+ change from baseline by study visit | Week 48
Proportion of virologic failures | Week 48
Incidence of adverse events, laboratory toxicities, and treatment discontinuations | Week 48
PK parameters: steady state (0-24hr) plasma AUC for emtricitabine; emtricitabine plasma trough concentration | Week 2 and between Weeks 8 to 24

CONTACTS AND LOCATIONS:
Locations (2):
- Romania (2):
  - Bucharest, Sector 2
  - Bucharest, Sector 3

REFERENCES:
- See also: Related Info — http://www.gilead.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/FTC-211_synopsis.pdf